CLINICAL TRIAL: NCT03459222
Title: A Phase 1/2 Study of Relatlimab (Anti-LAG-3 Monoclonal Antibody) Administered in Combination With Both Nivolumab (Anti-PD-1 Monoclonal Antibody) and BMS-986205 (IDO1 Inhibitor) or in Combination With Both Nivolumab and Ipilimumab (Anti-CTLA-4 Monoclonal Antibody) in Advanced Malignant Tumors
Brief Title: An Investigational Study of Immunotherapy Combinations in Participants With Solid Cancers That Are Advanced or Have Spread
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-048; 2018-000058-22 (EudraCT Number)
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Advanced Cancer
Keywords: Immunotherapy; Relatlimab; Nivolumab; Ipilimumab; BMS-986205
MeSH Terms: interventions — relatlimab; Nivolumab; linrodostat; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Relatlimab + Nivolumab + BMS-986205
  Interventions: Biological: Relatlimab; Biological: Nivolumab; Drug: BMS-986205
- Arm B (Experimental): Relatlimab + Nivolumab + Ipilimumab
  Interventions: Biological: Relatlimab; Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Relatlimab — Specified dose on specified days
  Other Names: BMS-986016
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
Drug: BMS-986205 — Specified dose on specified days
  Other Names: Linrodostat
  Arms: Arm A
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016
  Arms: Arm B

SUMMARY:
The purpose of this study is to demonstrate the safety and preliminary activity with triple combinations of relatlimab in combination with nivolumab and BMS-986205, or in combination with nivolumab and ipilimumab in immunotherapy-naive and pretreated populations across select advanced tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic confirmation of select incurable solid malignancies that are advanced (metastatic and/or unresectable), with measurable disease per RECIST v1.1
* Available tumor tissue for biomarker analysis
* Eastern Cooperative Oncology Group Performance Status (ECOG) status of 0 or 1

Exclusion Criteria:

* Known or suspected central nervous system (CNS) metastases or with the CNS as the only site of active disease
* History of interstitial lung disease / pneumonitis
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been cured, such as basal or squamous cell skin cancer
* Encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Number of clinical laboratory test abnormalities | Approximately 4 years
Number of Adverse Events (AEs) | Approximately 4 years
Number of Serious Adverse Events (SAEs) | Approximately 4 years
Number of AEs meeting protocol defined dose-limiting toxicity (DLT) criteria | Up to 6 weeks
Number of AEs leading to discontinuation | Approximately 4 years
Number of AEs leading to death | Approximately 4 years
Objective Response Rate (ORR) | Approximately 4 years
Disease Control Rate (DCR) | Approximately 4 years
Median Duration of Response (mDOR) | Approximately 4 years

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- United States (5):
  - Local Institution - 0006, Duarte, California
  - Local Institution - 0003, Aurora, Colorado
  - Local Institution - 0004, Baltimore, Maryland
  - Local Institution - 0005, St Louis, Missouri
  - Local Institution - 0001, Germantown, Tennessee
- Australia (2):
  - Local Institution - 0012, Wollstonecraft, New South Wales
  - Local Institution - 0011, Nedlands, Western Australia
- France (3):
  - Local Institution - 0017, Marseille
  - Local Institution - 0016, Toulouse
  - Local Institution - 0015, Villejuif
- Italy (3):
  - Local Institution - 0010, Forlì
  - Local Institution - 0009, Napoli
  - Local Institution - 0023, Rome
- Spain (5):
  - Local Institution - 0019, Barcelona
  - Local Institution - 0021, Madrid
  - Local Institution - 0018, Madrid
  - Local Institution - 0022, Málaga
  - Local Institution - 0020, Pamplona
- Switzerland (2):
  - Local Institution - 0008, Lausanne
  - Local Institution - 0007, Zurich
- United Kingdom (2):
  - Local Institution - 0013, Headington
  - Local Institution - 0014, Newcastle upon Tyne

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com